CLINICAL TRIAL: NCT00159159
Title: LOW CYCLO: A Multicenter, Prospective, Randomized Study Evaluating the Benefit, on Renal Function, of Two Doses of Ciclosporine: Low Dose Versus Usual Dose, in Association With Mycophenolate and Corticoïds, in de Novo Cardiac Transplant
Brief Title: LOW CYCLO: Study Evaluating the Benefit of Two Doses of Ciclosporine in de Novo Cardiac Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2003.325
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Cardiac Transplantion
Keywords: Cardiac Transplant; ciclosporine; immunosuppressive
MeSH Terms: interventions — Cyclosporins

INTERVENTIONS:
Drug: Ciclosporine 130 µg/l < T0 ciclosporinemia < 200 µg/l
Drug: Ciclosporine 200 µg/l < T0 ciclosporinemia < 300 µg/l

SUMMARY:
Primary Objective:

* Evaluation of the benefit on renal function of one year of a low dose of ciclosporine versus the usual dose

Secondary Objective:

* To evaluate the immunosuppressive efficacy and tolerance of the treatment

Study Duration:

Twelve months for each patient

Study Treatment: Ciclosporine

Group A: low dose >= 130 µg/l < T0 ciclosporinemia < 200 µg/l; Group B: standard dose >= 200 µg/l < T0 ciclosporinemia < 300 µg/l.

Study Visits:

One visit every 15 days, for the first three months; then 1 visit every month, for 6 months; and 1 visit at 9 and 12 months.

Associated Treatments:

* Mycophenolate (Cellcept®), 3g a day
* Corticoids, as used for transplanted patients

Randomization: Randomization will occur when it is decided that ciclosporine will be introduced.

ELIGIBILITY:
Inclusion Criteria:

Recipient:

* Males or females, ages > 18 < 65.
* First cardiac transplant.
* Negative pregnancy test for females of childbearing potential, at screening. Efficient method of contraception must be used during the study.
* Written informed consent.

Donor:

* Cold ischemia duration < 6 hours

Exclusion Criteria:

Recipient:

* Unstable hemodynamic status at randomization.
* Patient with assisted circulation, considered unstable.
* Serum creatinine > 250 µmol/l.
* Nursing or pregnant females.
* HIV positive.
* PCR hepatitis C virus (HCV) positive or hepatitis B surface (Hbs) antigen positive (within 6 months prior to study).
* Multi-organ graft or retransplant.
* History of cancer (evolving, or within 5 years, except for epidermoid or basocellular localised cutaneous carcinoma).
* Use of any investigational product and/or participation in another clinical research study within the last 30 days prior to study entry.
* Any substance abuse or any psychiatric disorder
* Contra-indication to study treatments.
* Unable to introduce ciclosporine within 4 days after transplant.

Donor:

* Known coronary pathology or cardiac disease.
* HBsAg positive or HCV positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106
Dates: Start 2004-03

PRIMARY OUTCOMES:
Evolution of renal function, as assessed by the evolution between the two treatment groups at 12 months versus baseline serum creatinine level

SECONDARY OUTCOMES:
Area under curve of creatinine at 12 months
Cystatin C level at 1, 2, 3, 6 and 12 months
Creatinine clearance at 6 and 12 months
Proteinuria and microalbuminuria at 6 and 12 months
Secondary outcomes include those linked to the immunosuppressive efficacy and tolerance of the treatment: Difference in appearance incidence of acute graft reject and adverse events
Myocardial biopsy (International Society of Heart and Lung Transplantation [ISHLT] grades)
Difference in the evolution of left ventricular function and cardiovascular risk factors between the two groups at 6 and 12 months versus baseline: left ventricular ejection fraction and shortening fraction (echocardiogram)
systolic and diastolic blood pressure
fasting glycemia, total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Pascale BOISSONNAT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Pascale BOISSONNAT, Lyon, France

REFERENCES:
- [Derived] Boissonnat P, Gaillard S, Mercier C, Redonnet M, Lelong B, Mattei MF, Mouly-Bandini A, Pattier S, Sirinelli A, Epailly E, Varnous S, Billes MA, Sebbag L, Ecochard R, Cornu C, Gueyffier F. Impact of the early reduction of cyclosporine on renal function in heart transplant patients: a French randomised controlled trial. Trials. 2012 Dec 3;13:231. doi: 10.1186/1745-6215-13-231. PMID 23206408